CLINICAL TRIAL: NCT03601702
Title: Multicentric Observational Prospective Study on the Use of the EmboTrap ® II Revascularization Device (Neuravi) in Acute Ischemic Stroke
Brief Title: EmboTrap ® II Revascularization Device (Neuravi) in Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Niguarda Hospital (Other)
Collaborators: Neuravi Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: REGISTRAP
Record Dates: First submitted 2018-05-11; First posted 2018-07-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; endovascular treatment; stent retriever device; mechanical thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EmboTrap ® II Device: The study group consists of the patients with acute ischemic stroke from large vessel occlusion treated with EmboTrap ® II Device (Neuravi)
  Interventions: Device: Mechanical thrombectomy with EmboTrap ® II Device

INTERVENTIONS:
Device: Mechanical thrombectomy with EmboTrap ® II Device — Endovascular treatment with mechanical thrombectomy using EmboTrap ® II Device (Neuravi)

SUMMARY:
The primary aim of Registrap study is to assess the safety and effectiveness of the EmboTrap®II Clot Retriever device (Neuravi) in patients with acute ischemic stroke from large vessel occlusion.

DETAILED DESCRIPTION:
Registrap is a prospective, single-arm, multicenter, observational registry of the Embotrap®II Clot Retriever (NEURAVI) open to any Neurointerventional Department in Europe with experience in mechanical thrombectomy with the EmboTrap® II device Clot Retriever (5 cases already done) and a number of stroke procedures/year greater than 30.

The EmboTrap®II Clot Retriever (Neuravi) is CE-marked and represents one of the possible treatment devices, chosen by physicians according to their experience and practice, in acute ischemic stroke treatment.

Being REGISTRAP an observational registry and considering that different approaches and devices are available on the market, the investigators are aware that operators' preferences could represent a selection bias. The Screening Log will collect all the stroke cases treated from each centre during the enrollment period to show the rate of EmboTrap®II Clot Retriever (Neuravi) use over the total cases treated and the reasons for choosing other devices. The registry will enroll at least 100 consecutive patients presenting within 12 hours from symptom onset with a Large Vessel Occlusion (LVO) on CTA or MRA in the Anterior or Posterior Proximal Cerebral Vasculature up to A1, M1, Dominant M2, P1 who will be treated using the EmboTrap®II Clot Retriever (Neuravi) as first intention and used according to the Instructions For Use. The registry objectives are to evaluate the efficacy/safety of the device Embotrap II Clot Retriever(Neuravi), as first line treatment in the restoration of cerebral blood flow in cases of acute ischemic stroke from Large Vessel Occlusion. Efficacy is considered when a "modified Treatment in Cerebral Infarction" (mTICI) score of 2b or greater is achieved in the vessel treated with the (Neuravi). Safety refers to the rate of procedure-related and device-related hemorrhages. Number and severity of hemorrhages will be evaluated considering site and size. The first follow-up control will occur at 1 to 10 days post-procedure, the second at 90 days+/-14 days. In addition to the sample, the patients meeting the inclusion criteria and treated using the EmboTrap®II Clot Retriever (Neuravi) as second intention, will also be included in the study and considered only for a specific secondary endpoint.

ELIGIBILITY:
Inclusion Criteria

* Signed Informed Consent Form
* Large Vessel Occlusion on CTA or MRA in the Anterior or Posterior Proximal Cerebral Vasculature up to A1, M1, Dominant M2, P1
* ASPECTS ≥ 6
* Mismatch or good collaterals showed at MR or multiphasic CTA or pCT
* Groin Puncture performed within 12 hours from symptom onset
* Use of EmboTrap® II Revascularization Device (Neuravi) as the first or second line treatment

Exclusion criteria

* Informed consent not given
* Extracranial or tandem occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry enrolls acute ischemic stroke patients presenting within 12 hours from neurological symptom onset with a Large Vessel Occlusion (LVO) on CTA or MRA in the Anterior or Posterior Proximal Cerebral Vasculature up to A1, M1, Dominant M2, P1 who will be treated using the EmboTrap®II Clot Retriever (Neuravi) according to the Instructions For Use
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety: device -related haemorrhages rate showed by CT/MR | 10 days
  Procedure-related mortality rate
Efficacy: Restoration of cerebral blood flow at the end of the procedure | 1 day
  Restoration of cerebral blood flow

SECONDARY OUTCOMES:
Rate of embolisation in new territories | 10 days
  Rate of embolisation in new territories
Restoration of cerebral flow to achieve mTICI 2b/3 as second line treatment | 1 day
  Efficacy of the device Embotrap II Clot Retriever (Neuravi), as second line treatment in the restoration of cerebral flow to achieve mTICI 2b/3

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Investigators' meeting
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Each six months
URL: http://www.registrap.org